CLINICAL TRIAL: NCT03876535
Title: A Performance Evaluation of the Nanomix eLab® C-Reactive Protein, Procalcitonin, and Lactate Assays With the Nanomix eLab System
Brief Title: Performance Evaluation of the Nanomix eLab® CRP, PCT, and LAC Assays With the Nanomix eLab System
Status: Completed | Type: Observational
Sponsor: Nanomix (Industry)
Responsible Party: Sponsor
Other Study IDs: Nanomix-010s
Record Dates: First submitted 2019-03-12; First posted 2019-03-15 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2019-09

CONDITIONS: Sepsis; SIRS
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma samples (without cells/ RNA/DNA) will be aliquoted and stored at Sponsor for future analysis/ projects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Nanomix eLab® System molecular diagnostic test (non-interventional) — This is not an interventional study. It involves performance equivalence demonstration of a point of care diagnostic system to FDA cleared predicate devices currently used in sepsis and SIRS diagnosis.

SUMMARY:
The performance of the eLab C-Reactive Protein, Procalcitonin, and Lactate Assays will be demonstrated during a method comparison study in which venous whole blood and plasma samples are used. eLab results will be compared to an FDA cleared predicate device. Demographic information will be collected for the subject. Venous blood will be collected in 2 Li-heparinized tubes (2-4ml per tube). One tube will be used for testing at the site and the second tube will be processed to plasma for storage and subsequent shipment to a designated testing site. Whole blood samples will be tested on the eLab C-Reactive Protein, Procalcitonin, and Lactate test as soon as possible after collection; testing on whole blood must be completed within 30 minutes of collection. A predicate Lactate test will also be run as soon as possible after collection; testing of WB on the predicate must be completed within 30 minutes of collection. Plasma will be separated from the whole blood via centrifugation within 30 minutes of collection and tested on the eLab C-Reactive Protein, Procalcitonin, and Lactate Assays and started on predicate CRP and PCT devices (If available at the site) within 30 minutes of the eLab whole blood test. The remainder of the plasma specimen and plasma from the second collection tube will be frozen within one hour of collection, then stored at approximately -20 degrees C or colder.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older
* Must have provided written informed consent
* Admitted to ICU, Emergency Department or other medical wards for acute illness and observation of infection and meeting SIRS criteria (such as elevated heart rate, tachypnea, hypotension, fever, hypothermia, or elevated respiratory rate)

Exclusion Criteria:

* Pregnant or nursing
* Admitted to ICU after trauma
* Admitted to ICU after surgery
* Cardiogenic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteers from medical wards presenting with acute illness, observation of infection and meeting SIRS criteria.
Sampling Method: Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Estimates of bias relative to an FDA cleared predicate device using CLSI EP9-A3 as a guideline. | One timepoint at enrollment
  An analysis of the results from 150-200 subjects collected across the three (3) sites will be performed to accomplish the analytical comparison endpoints. If the analysis requires more samples to cover the assay range, then, the study may be continued and more subjects enrolled. A minimum of 25 percent of the samples must have values near the clinical significant concentration. In order to meet this requirement up to 10 % of samples may be spiked. Clinical significant concentrations for CRP are defined as values greater than 10 mg/L; PCT values greater than 0.5 ng/mL and LAC values greater than 2 mmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Landess, Study Director — Nanomix
Locations (1):
- UCSF- San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No